CLINICAL TRIAL: NCT02140164
Title: Pilot Study to Evaluate Oral Minocycline in the Treatment of Cystoid Macular Edema Associated With Retinitis Pigmentosa
Brief Title: Study of Oral Minocycline in Treating Bilateral Cystoid Macular Edema Associated With Retinitis Pigmentosa
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Collaborators: The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 140108; 14-EI-0108 (Other: NIH Combined NeuroScience Institutional Review Board)
Record Dates: First submitted 2014-05-14; First posted 2014-05-16 (Estimated); Results first posted 2017-01-16 (Estimated); Last update posted 2024-04-17 (Actual); Status verified 2017-11

CONDITIONS: Retinitis Pigmentosa
Keywords: Cystoid Macular Edema; Minocycline; Microglia; Retinitis Pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa; Macular Edema; cyclopia sequence | interventions — Minocycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Minocycline (Experimental): Oral administration of minocycline
  Interventions: Drug: Minocycline

INTERVENTIONS:
Drug: Minocycline — Oral dose of 100 mg (or appropriate weight-adjusted pediatric dose) of minocycline twice daily for 12 months.
  Other Names: Dynacin; serial number 73419626; Minocin; serial number 72309825; Minocin PAC; Myrac; serial number 76589055; Solodyn; serial number 78883462; Vectrin; serial number 78188505

SUMMARY:
Background:

- Some people with retinitis pigmentosa (RP) have macular edema (swelling) in the central retina. This can cause decreased central vision. The cause of macular edema is unknown, but may involve inflammation. The drug minocycline might help prevent inflammation and therefore might help treat macular edema and improve central visual function .

Objectives:

- To see if minocycline helps people with RP and macular edema.

Eligibility:

- People 12 years and older with RP who have macular edema in at least on eye.

Design:

* Participants will be screened with medical and eye disease history. They will have an eye exam and blood tests. One eye with macular edema will be the study eye. If both eyes are affected, one will be designated the study eye.
* Participants will visit the clinic at least 9 times over at least 14 months. The first 3 study visits will be monthly, then every 2 months.
* Participants will start taking minocycline after visit 3. They will take 1 pill twice daily for at least 1 year.
* Participants will keep a medicine diary and bring it to each visit with their pill bottle and unused pills.

At each study visit, participants will have some or all of the following tests:

* eye and thyroid exams
* blood and pregnancy tests
* microperimetry: participants will press a button when they see a light on a computer screen
* visual field measurement: participants will look at spots on a white screen to test side vision
* electroretinogram: A person will be dark adapted by sitting in the dark for 30 minutes. After the placement of numbing eye drops, special contact lenses will be placed . The participant will watch flashing lights and recordings will be made.

DETAILED DESCRIPTION:
Objective:

Retinitis pigmentosa (RP) is a broad category of genetically heterogeneous diseases involving progressive visual loss by a constriction of visual field and loss of night vision. In up to one-third of patients, the peripheral vision loss can be compounded by central visual acuity loss from the development of cystic macular changes. While RP is a genetic disease, the etiology of progressive cell death, including that of associated cystoid macular edema (CME), is not completely understood. Inflammatory processes involving the activation of resident immune cells of the retina called microglia have been hypothesized to contribute. Minocycline inhibits the activation of microglia, decreasing the production of inflammatory factors implicated in RP progression. The objective of this study is to investigate the safety and possible efficacy of oral minocycline in participants with CME and RP.

Study Population:

Five participants, ages 12 and older, with unilateral or bilateral CME associated with RP will be enrolled initially. However, up to an additional five participants may be enrolled to replace participants who may withdraw from the study prior to reaching the Month 6 visit.

Design:

This is a pilot, single-center, uncontrolled, open-label, prospective, Phase 1/2 clinical trial to evaluate minocycline as a potential treatment for CME secondary to RP. A pre-treatment phase lasting two months will be instituted prior to investigational product (IP) initiation to assess the anatomical variability of CME as well as variability of other measurable parameters as part of the natural history of the disease. Participants will receive an oral dose of 100 mg (or appropriate weight adjusted pediatric dose) of minocycline twice daily for 12 months. There will be a common termination date, which will take place when the last recruited participant has received 12 months of IP. Participants who were recruited in the earlier part of the study will continue taking IP and be followed every two months until the common termination date. At each visit, participants will have visual acuity measured and will undergo optical coherence tomography (OCT) testing to measure retinal thickness. Measures of central visual field sensitivity full-field electroretinograms (ERG) and microperimetry (MP-1) will also be collected.

Outcome Measures:

The primary outcome is the change in CME based on OCT measurements in the study eye at 6 months compared to pre-treatment values. Secondary outcomes include changes in OCT thickness, changes in amplitude of photopic and scotopic responses on ERG testing, changes in microperimetry, and changes in visual field as measured by HVF 30-2 visual field testing at 6 months and 12 months compared to pre-treatment values, as well as CME changes on OCT at 12 months compared to pre-treatment values. Pre-treatment measurements will be analyzed to measure the natural variability of the CME as well as to measure the variability of the functional testing. Safety outcomes will include the number and severity of adverse events (AEs). Ocular safety outcomes will be indicated by changes in visual acuity, ocular surface changes, intraocular inflammation and any other ocular changes not consistent with the natural progression of RP.

ELIGIBILITY:
* INCLUSION CRITERIA:
* To be eligible, the following inclusion criteria must be met, where applicable.
* Participant must be 12 years of age or older.
* Participant (or legal guardian) must understand and sign the protocol's informed consent document.
* Participant must have evidence of retinitis pigmentosa (RP) as defined by characteristic electroretinogram (ERG) responses and visual fields.
* Participant must be able to swallow pills.
* Participant must have normal renal function and liver function or have mild abnormalities not above grade 1 as defined by the Common Terminology Criteria for Adverse Events v4.0 (CTCAE).
* Participant must agree to minimize exposure to sunlight or artificial ultraviolet (UV) rays and to wear protective clothing, sunglasses and sunscreen [minimum sun protection factor (SPF) 15] if s/he must be out in the sun.
* Any female participant of childbearing potential must have a negative pregnancy test at screening and be willing to undergo pregnancy tests throughout the study.
* Any female participant of childbearing potential and any male participant able to father children must have (or have a partner who has) had a hysterectomy or vasectomy, be completely abstinent from intercourse or must agree to practice two acceptable methods of contraception throughout the course of the study and for at least one week after investigational product (IP) discontinuation. Acceptable methods of contraception include:

  * hormonal contraception (i.e., birth control pills, injected hormones, dermal patch or vaginal ring),
  * intrauterine device,
  * barrier methods (diaphragm, condom) with spermicide, or
  * surgical sterilization (hysterectomy or tubal ligation).

EXCLUSION CRITERIA:

A participant is not eligible if any of the following exclusion criteria are present.

* Participant is actively receiving study therapy in another investigational study.
* Participant is started on (or changed dosage of) topical or systemic carbonic anhydrase inhibitor (CAI) treatment in the 3 months prior to enrollment.
* Participant is actively receiving systemic steroids or has received systemic steroids in the 3 months prior to enrollment.
* Any female participant of childbearing potential that is pregnant, breast-feeding or planning to become pregnant during the study.
* Participant is expected to be unable to comply with study procedures or follow-up visits.
* Participant has evidence of an ocular disease other than RP in either eye that may confound the outcome of the study (e.g., diabetic retinopathy with 10 or more hemorrhages or microaneurysms, uveitis, pseudovitelliform macular degeneration, severe myopia).
* Participant is on ocular or systemic medications known to be toxic to the lens, retina or optic nerve (e.g., ethambutol, chloroquine, or hydroxychloroquine).
* Participant has a condition that would preclude participation in the study (e.g., unstable medical status including blood pressure and glycemic control) by interfering with the participant s ability to engage in the required protocol evaluation and testing and/or comply with study visits.
* Participant has a history of chronic renal failure requiring dialysis or kidney transplant.
* Participant has a history of chronic hepatitis or liver failure.
* Participant has a history of thyroid cancer.
* Participant has an allergy or hypersensitivity to minocycline or any drug in the tetracycline family.
* Participant is currently taking a tetracycline medication.
* Participant is taking any medication that could adversely interact with minocycline such as methoxyflurane.
* Participant has a prior history of idiopathic intracranial hypertension.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-05; Primary Completion 2015-11 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine A Cukras, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boughman JA, Conneally PM, Nance WE. Population genetic studies of retinitis pigmentosa. Am J Hum Genet. 1980 Mar;32(2):223-35. PMID 7386458
- [Background] Li ZY, Possin DE, Milam AH. Histopathology of bone spicule pigmentation in retinitis pigmentosa. Ophthalmology. 1995 May;102(5):805-16. doi: 10.1016/s0161-6420(95)30953-0. PMID 7777280
- [Background] Chang GQ, Hao Y, Wong F. Apoptosis: final common pathway of photoreceptor death in rd, rds, and rhodopsin mutant mice. Neuron. 1993 Oct;11(4):595-605. doi: 10.1016/0896-6273(93)90072-y. PMID 8398150
- [Result] Dave AD, Chen KG, Chiang TT, Singaravelu J, Alvarez JA, Wong WT, Cukras CA. Oral minocycline for the treatment of retinitis pigmentosa-associated cystoid macular edema: results of a phase I/II clinical trial. Graefes Arch Clin Exp Ophthalmol. 2023 Aug;261(8):2209-2220. doi: 10.1007/s00417-023-05986-6. Epub 2023 Mar 8. PMID 36882562
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-EI-0108.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Five participants, ages 12 and older, with cystoid macular edema (CME) secondary to retinitis pigmentosa (RP) who meet the eligibility criteria will be initially accrued; however, up to an additional five participants may be enrolled to replace participants who may withdraw from the study prior to reaching Month 6
Period: Overall Study
Arm/Group | Minocycline
Started | 7
Completed | 5
Not Completed | 2
Not completed — Cystoid Macular Edema (CME) resolved | 2

BASELINE CHARACTERISTICS:
Arm/Group | Minocycline
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.7 (8.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Cystoid Macular Edema (CME) Based on Optical Coherence Tomography (OCT) Measurements in the Study Eye at 6 Months Compared to the Average of the Pre-treatment Values.
Description: Three visits (two pre-treatment and one baseline) were conducted prior to the receipt of investigational product (IP) and an average of the OCT measurements at these three visits was used as the pre-treatment value.
Time Frame: Pre-treatment and 6 Months
Population: Participants receiving investigational product (IP) at the Month 6 visit were included in the primary efficacy analysis.
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Minocycline
Number analyzed (Participants) | 5
microns | -16.7 (42.16)

2. Secondary Outcome: Change in Cystoid Macular Edema (CME) Based on Optical Coherence Tomography (OCT) Measurements in the Study Eye at 12 Months Compared to the Average of the Pre-treatment Values
Description: as for outcome 1
Time Frame: Pre-treatment and 12 Months
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Minocycline
Number analyzed (Participants) | 5
microns | -37.3 (52.90)

3. Secondary Outcome: Changes in Amplitude of Photopic and Scotopic Responses on Electroretinogram (ERG) Testing at 6 Months as Compared to the Average of Pre-treatment Values
Description: This outcome measure will not be reported.
Time Frame: Pre-Treatment and 6 Months
Population: Participants had non-recordable ERGs; therefore, changes could not be measured.
Arm/Group | Minocycline
Number analyzed (Participants) | 0

4. Secondary Outcome: Changes in Amplitude of Photopic and Scotopic Responses on Electroretinogram (ERG) Testing at 12 Months as Compared to the Average of Pre-treatment Values
Description: This outcome measure will not be reported.
Time Frame: Pre-treatment and 12 Months
Population: Participants had non-recordable ERGs; therefore, changes could not be measured.
Arm/Group | Minocycline
Number analyzed (Participants) | 0

5. Secondary Outcome: Change in Microperimetry at 6 Months as Compared to the Average of Pre-treatment Values
Description: Three visits (two pre-treatment and one baseline) were conducted prior to the receipt of investigational product (IP) and an average of the microperimetry measurements at these three visits was used as the pre-treatment value.
Time Frame: Pre-treatment and 6 Months
Measure: Mean (Standard Deviation); unit: decibels (dB)
Arm/Group | Minocycline
Number analyzed (Participants) | 5
decibels (dB) | -1.01 (0.36)

6. Secondary Outcome: Change in Microperimetry at 12 Months as Compared to the Average of Pre-treatment Values
Description: as for outcome 5
Time Frame: Pre-treatment and 12 Months
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Minocycline
Number analyzed (Participants) | 5
dB | -1.02 (0.45)

7. Secondary Outcome: Change in Visual Field as Measured by HVF 30-2 Visual Field Testing at 6 Months as Compared to the Average of Pre-treatment Values
Description: Three visits (two pre-treatment and one baseline) were conducted prior to the receipt of investigational product (IP) and an average of the HVF 30-2 measurements at these three visits was used as the pre-treatment value.
Time Frame: Pre-treatment and 6 Months
Population: Two participants had to switch to HVF 10-2; therefore they were not included in the analysis.
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Minocycline
Number analyzed (Participants) | 3
dB | -3.62 (5.80)

8. Secondary Outcome: Change in Visual Field as Measured by HVF 30-2 Visual Field Testing at 12 Months as Compared to the Average of Pre-treatment Values
Description: as for outcome 7
Time Frame: Pre-treatment and 12 Months
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Minocycline
Number analyzed (Participants) | 3
dB | 1.69 (5.52)

9. Secondary Outcome: Number of Study Eyes Achieving a 15-letter or More Worsening in Electronic Visual Acuity (EVA) at 12 Months as Compared to Baseline
Description: Visual Acuity was measured by a certified tester using an electronic visual acuity testing machine based on the Early Treatment Diabetic Retinopathy Study (ETDRS) method.
Time Frame: Baseline and 12 Months
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Minocycline
Number analyzed (Participants) | 5
Number analyzed (eyes) | 5
eyes | 0

10. Secondary Outcome: Number of Ocular Adverse Events
Time Frame: Study Duration, up to 16 Months
Population: All participants were included in the safety analysis.
Measure: Number; unit: adverse events
Arm/Group | Minocycline
Number analyzed (Participants) | 7
adverse events | 3

11. Secondary Outcome: Number of Non-ocular Adverse Events
Time Frame: Study Duration, up to 16 Months
Population: All participants were included in the safety analysis.
Measure: Number; unit: adverse events
Arm/Group | Minocycline
Number analyzed (Participants) | 7
adverse events | 12

12. Secondary Outcome: Number of Severe Adverse Events
Time Frame: Study Duration, up to 16 Months
Population: All participants were included in the safety analysis.
Measure: Number; unit: adverse events
Arm/Group | Minocycline
Number analyzed (Participants) | 7
adverse events | 0

ADVERSE EVENTS:
Time Frame: Study Duration, up to 16 months
Description: Adverse events were collected on and after the baseline visit, and when investigational product (IP) began.
Arm/Group | Minocycline
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 6/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Minocycline (N=7)
Nasopharyngitis (Infections and infestations) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Visual acuity reduced (Eye disorders) | 1 (2)
Blood potassium increased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes